CLINICAL TRIAL: NCT05938322
Title: Compliance With Ketogenic Diet in Patients Undergoing Radiotherapy for Pelvic Cancers: a Prospective, Randomized, Mono-centric Study
Brief Title: Ketogenic Diet Compliance in Patients Undergoing Radiotherapy for Pelvic Cancers
Acronym: KOMPARC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Mele Maria Cristina, Prof., Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 5812
Record Dates: First submitted 2023-06-12; First posted 2023-07-10 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Rectal Cancer
Keywords: Rectal Cancer; Ketogenic Diet
MeSH Terms: conditions — Rectal Neoplasms | interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketogenic Diet (Experimental): In the group of intervention is prescribed a ketogenic diet plan.
  Interventions: Other: Ketogenic Diet
- Standard Diet (Active Comparator): The control group (SD) will follow the Mediterranean diet pattern based on ESPEN (European Society of Parenteral and Enteral Nutrition) guidelines
  Interventions: Other: Standard Diet

INTERVENTIONS:
Other: Ketogenic Diet — In the group of intervention is prescribed a ketogenic diet plan characterized by the following composition: carbohydrates < 30g/day, 1.2g-1.5g protein/kg/day and lipids > 65%.
  This diet will be followed during the period of treatment with chemo-radiotherapy (5 weeks)
  Arms: Ketogenic Diet
Other: Standard Diet — The control group (SD) will follow the Mediterranean diet pattern based on ESPEN guidelines (carbohydrates 45-55%, protein 15-20% and lipids 30-35%).
  Arms: Standard Diet

SUMMARY:
Patients with locally advanced non-metastatic adenocarcinoma of the rectum undergoing chemoradiation therapy will be assigned to 2 groups:

* the intervention group will be prescribed an individualized ketogenic eating plan to be followed throughout the treatment period
* the control group will be prescribed a diet therapy plan treatment following the international guidelines of clinical nutrition, also to be followed during treatment

DETAILED DESCRIPTION:
Some days before the start of radiotherapy there will be the first visit in which patients will be enrolled and placed in one of the following two groups:

* The intervention group (KD) will be prescribed a ketogenic diet therapy plan characterized by the following composition: carbohydrates < 30g/day, 1.2g-1.5g protein/kg/day and lipids > 65%.
* The control group (SD) will be prescribed a nutrition plan based on the Mediterranean diet model according to ESPEN guidelines (carbohydrates 45-55%, protein 15-20% and lipids 30-35%) There will then be two additional follow-ups for patients: one during the period of therapy and one at the end of therapy.

Compliance with diet therapy treatment (SD vs. KD) will be assessed by analysis of a food diary that the patient will be asked to complete.

During follow-ups it will be assessed:

* BMI and body composition (by bioimpedance analysis)
* Muscle strength and physical performance (by hand grip test and sit-to-stand test) Compliance with and toxicity of radiochemotherapy treatment will be assessed at the radiochemotherapy visits (3 visits during treatment)

ELIGIBILITY:
Inclusion Criteria:

* Histologic confirmation of rectal adenocarcinoma
* Locally advanced rectal cancer
* Patients undergoing neoadjuvant radiotherapy treatment
* Signature of informed consent to the processing of personal data

Exclusion Criteria:

* Severely malnourished patients according to GLIM (Global Leadership Initiative on Malnutrition) criteria
* Patients treated for palliative purposes
* Patients with metastatic disease
* Diabetes mellitus
* Pregnancy or lactation
* Significant food allergies that would make the person unable to consume the food provided
* Refusal to participate in the proposed clinical trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Adherence to the ketogenic diet | 2 months
  The primary objective is to assess the adherence to the diet therapy treatment plan (SD vs. KD). It will be verified through a food diary that will be given to the patient during the first visit.
  The patients will fill out the questionnaire and return it at future visits.

SECONDARY OUTCOMES:
Assessment of fat mass (FM) in the group of patients on ketogenic diet (KD) compared with the control group | 2 months
  The assessment will be carried out through the use of an impedance analysis (BIA)
Evaluation of maintenance of metabolically active mass (BCM) in the group of patients on ketogenic diet (KD) compared with the control group | 2 months
  The assessment will be carried out through the use of an impedance analysis (BIA)
Investigate the impact of BCM maintenance on metabolic, inflammatory, hematologic and endocrine response | 2 months
  The assessment will be carried out through blood test analysis
Evaluation of the correlation between ketogenic diet (KD) and metabolic, inflammatory, hematologic and endocrine response | 2 months
  The assessment will be carried out through blood test analysis
Evaluation of the tolerability to the treatment | 2 months
  Radiotherapy interruptions will be evaluated
Evaluation of the response to the treatment | 2 months
  The assessment will be carried out through pelvic MRI analysis, clinical evaluation, and pathological response
Investigate indices of quality of life | 2 months
  Investigating patients' quality of life through questionnaires administered at the beginning and at the end of treatments. The questionnaires used are EORT ( European Organisation for Research and Treatment of Cancer) QLQ (quality of life questionnaire)-30, QLQ - CR29 and CAX-24 (cancer cachexia-specific questionnaire), and PRT-20 (quality of life questionnaire for proctitis).

CONTACTS AND LOCATIONS:
Overall Officials: Maria Cristina Mele, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli, IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: No